CLINICAL TRIAL: NCT03636204
Title: A First in Human Phase 1 Study in Healthy Volunteers and in Participants With Frontotemporal Dementia (FTD) With Granulin Mutation
Brief Title: A First in Human Study in Healthy Volunteers and in Participants With Frontotemporal Dementia With Granulin (GRN) Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alector Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL001-1
Record Dates: First submitted 2018-07-12; First posted 2018-08-17 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Healthy; Frontotemporal Dementia
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AL001 (Experimental): Up to six single ascending doses of AL001
  Interventions: Biological: AL001
- Saline Solution (Placebo Comparator): Saline solution will be administered as a single infusion for each cohort in a ratio of 6 active and 2 placebo subjects
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AL001 — Active dose of AL001
  Arms: AL001
Other: Placebo — Saline solution administered as a single infusion as palcebo.
  Arms: Saline Solution

SUMMARY:
A first in human phase 1 study in healthy volunteers and participants with Granulin (GRN) mutation causative of frontotemporal dementia (FTD) to assess AL001 safety, tolerability, pharmacokinetics, and pharmacodynamics

DETAILED DESCRIPTION:
This is a first-in-human Phase 1 study designed to investigate the safety, tolerability, PK and PD of intravenously administered AL001 in Healthy Volunteers and FTD-GRN mutation carriers.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.0-35.0 kg/m2
* 45-120 kg, inclusive
* At screening, females must be non-pregnant and non-lactating, or of nonchildbearing potential (either surgically sterilized or physiologically incapable of becoming pregnant, or at least 1-year postmenopausal (amenorrhoea duration of 12 consecutive months); nonpregnancy will be confirmed for all females by a pregnancy test conducted at screening, (each) admission, and at follow-up.
* Female participants of child-bearing potential must agree to use adequate contraception from screening until 90 days after the follow-up visit.
* In good physical health on the basis of no clinically significant findings from medical history, physical examination (PE), laboratory tests, 12 lead ECG, and vital signs, as judged by the Investigator.
* Willingness and able to comply with the study protocol, in the investigator's judgement.

Exclusion Criteria:

* Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins.
* Positive drug or alcohol at screening and prior to first dose
* History of alcohol abuse or substance abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability of AL001 measured by number of subjects with adverse events and Dose Limiting Adverse Event (DLAEs) | 85 days
  Incidence of adverse events and dose limiting Adverse Events during the DLAE observation period and/or study treatment periods.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of AL001 | 85 days
  Serum and cerebrospinal fluid (CSF) concentration of AL001 at specified time points
Maximum plasma concentration (Cmax) for AL001 | 85 days
  Evaluate Cmax for serum and CSF concentration of AL001 at specified time points
Area under the curve concentration (AUC) for AL001 | 85 days
  Evaluate AUC for serum and CSF concentration of AL001 at specified time points

CONTACTS AND LOCATIONS:
Overall Officials: George Stoica, Principal Investigator — Bioclinica Research
Locations (8):
- United States (5):
  - University of Alabama, Birmingham, Alabama
  - UCSF, San Francisco, California
  - Study site, Orlando, Florida
  - Mayo Clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Canada (2):
  - Lawson Health Research Institute, St. Joseph's, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto
- University College London, London, United Kingdom

REFERENCES:
- [Derived] Kurnellas M, Mitra A, Schwabe T, Paul R, Arrant AE, Roberson ED, Ward M, Yeh F, Long H, Rosenthal A. Latozinemab, a novel progranulin-elevating therapy for frontotemporal dementia. J Transl Med. 2023 Jun 15;21(1):387. doi: 10.1186/s12967-023-04251-y. PMID 37322482